CLINICAL TRIAL: NCT03689400
Title: Changes of Pain and Functional Parameters in Back Pain Patients With or Without Radiculopathy Over Time
Brief Title: Changes of Pain and Functional Parameters in Back Pain Patients Over Time
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Collaborators: Cantonal Hospital Graubuenden (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00637_KSGR
Record Dates: First submitted 2018-08-29; First posted 2018-09-28 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Changes Over Time in Pain and Functional Parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Back pain affects patients' daily life. Patients can suffer from various symptoms which appear intermittent or permanent; pain, sensory malfunction, reduction of muscular strength and coordination. Therefore, patients are impaired in participation and activity.

Physiotherapy is recommended to improve those symptoms and to positively affect the cause of the problem. However, some patients do not benefit from physiotherapeutic treatment and require a surgery.

The investigators intend to attend patients suffering from back pain and to document the changes of pain and functional parameters over a period of 6 months. The investigators include pre-operative, post-operative or non-operated patients which allows to discuss the different treatment options and its effects.

DETAILED DESCRIPTION:
To assess pain and functional parameters physicians, medical staff and physiotherapist often use subjective clinical testings which impede the comparability of testings over time, between testers and between subjects.

Therefore, a second aim of this study is to evaluate each subjective clinical test with a standardized objective measurement tool.

ELIGIBILITY:
Inclusion Criteria:

* appointment at the neurosurgery department due to back pain
* German speaking
* willingness to see a physiotherapist
* willingness to participate in 3 measurements over 6 months

Exclusion Criteria:

* no appointment at the neurosurgery department due to back pain
* not German speaking
* no willingness to see a physiotherapist
* no willingness to participate in 3 measurements over 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators are looking for subjects suffering from back pain, who visit the neurosurgery department of the Cantonal hospital of Grisons in Chur to discuss the further treatment of their disease. The subjects get their normal medical and physiotherapeutical treatment independent of the study participation.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — SUPSI Landquart, Switzerland
Locations (1):
- Cantonal Hospital of Grisons, Chur, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bianchi G, Zweifel C, Hohenauer E, Santos JAR and Clijsen R (2025) Reliable outcome parameters in patients with lumbar radiculopathy attributed to disc herniation: an observational study. Front. Musculoskelet. Disord. 3:1672539. doi: 10.3389/fmscd.2025.1672539
- See also: Fulltext — https://www.frontiersin.org/journals/musculoskeletal-disorders/articles/10.3389/fmscd.2025.1672539/full

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Lumbar Disc Herniation Associated With Radiculopathy: Adult patients diagnosed with lumbar disc herniation associated with radiculopathy at the Cantonal Hospital of Graubünden. Physical assessment was done to diagnose LR; an MRI was performed to confirm the presence of an LDH. All patients included in this study received physiotherapy at the Cantonal Hospital Graubünden, regardless of whether they had undergone surgery beforehand.
Period: Overall Study
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Started | 19
Completed | 15
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Level of lesion [Count of Participants; unit: Participants]
  first sacral vertebra (S1) | 5
  fifth lumbar vertebra (L5) | 9
  fourth lumbar vertebra (L4) | 2
  third lumbar vertebra (L3) | 3
  second lumbar vertebra (L2) | 0
Side of lesion [Count of Participants; unit: Participants]
  Right | 9
  Left | 10
Type of treatment [Count of Participants; unit: Participants]
  Conservative only | 9
  Surgery and Conservative | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Visual Analog Scale Pain Scores
Description: Changes in pain were assessed using a unidimensional 10-cm Visual Analogue Scale. The scale ranged from one endpoint depicting a happy face, indicating "no pain," to the other endpoint depicting a sad face, indicating "worst possible pain." The distance in centimeters from the low end (0) of the VAS to the patient's mark was used as a numerical measure of pain severity. The lowest score was 0, indicating no pain, the maximum score 10, indicating worst possible pain. Higher scores indicate more severe pain.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Units on a scale
  Baseline | 3.6 (3.0)
  6 weeks follow-up | 1.2 (1.6)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 0.5 (1.3)

2. Primary Outcome: Changes in Visual Analog Scale Ratings of Numbness
Description: Changes in pain were assessed using a unidimensional 10-cm Visual Analogue Scale. The scale ranged from one endpoint depicting a happy face, indicating "no numbness," to the other endpoint depicting a sad face, indicating "worst possible numbness." The distance in centimeters from the low end of the VAS to the patient's mark was used as a numerical measure of pain severity. The lowest score was 0, indicating no numbness, the maximum score 10, indicating worst possible numbness. Higher scores indicate more severe numbness.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Units on a scale
  Baseline | 2.2 (2.3)
  6 weeks follow-up | 0.8 (1.8)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 0.3 (1.3)

3. Primary Outcome: Changes in Visual Analog Scale Ratings of Paresthesia
Description: Changes in pain were assessed using a unidimensional 10-cm Visual Analogue Scale. The scale ranged from one endpoint depicting a happy face, indicating "no paresthesia" to the other endpoint depicting a sad face, indicating "worst possible paresthesia." The distance in centimeters from the low end of the VAS to the patient's mark was used as a numerical measure of pain severity. The lowest score was 0, indicating no paresthesia, the maximum score 10, indicating worst possible paresthesia. Higher scores indicate more severe numbness.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Units on a scale
  Baseline | 3.3 (2.7)
  6 weeks follow-up | 0.9 (1.5)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 0.3 (1.3)

4. Primary Outcome: Changes in Anterior Flexion Measured in Centimeters
Description: The fingertip-to-floor (FTF) test (cm) was used to assess the lumbar maximal anterior flexion. Patients performed maximal flexion up to the pain threshold, keeping the elbows, fingers, and knees straight and the heels together.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Centimeter
  Baseline | 21.7 (16.3)
  6 weeks follow-up | 17.8 (14.9)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 11.8 (10.4)

5. Primary Outcome: Changes in Back Extension Measured in Degrees
Description: Extension was measured using a baseline bubble inclinometer. Patients performed maximal extension up to the pain threshold, keeping the elbows, fingers, and knees straight and the heels together.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Degree
  Baseline | 18.7 (8.0)
  6 weeks follow-up | 21.8 (5.8)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 27.9 (10.0)

6. Primary Outcome: Changes in Lateral Flexion Measured in Centimeters
Description: The fingertip-to-floor (FTF) test (cm) was used to assess the lumbar maximal lateral flexion. Patients performed maximal flexion up to the pain threshold, keeping the elbows, fingers, and knees straight and the heels together. The contralateral hip remained in contact with the treatment table during lateral flexion.
Time Frame: Baseline, 6 weeks, 6 months
Population: four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Centimeter
  right side: Basline | 51.3 (4.4)
  right side: 6 weeks follow-up | 49.9 (4.0)
  right side: 6 months follow-up: number analyzed (Participants) | 15
  right side: 6 months follow-up | 49.2 (4.4)
  Left side: Baseline | 50.2 (5.4)
  Left Side: 6 weeks follow-up | 49.4 (3.5)
  Left side: 6 months follow-up: number analyzed (Participants) | 15
  Left side: 6 months follow-up | 48.6 (3.7)

7. Primary Outcome: Changes in the Maximal Isometric Strength in Newton
Description: Maximal isometric strength was tested using the NOD hand-held dynamometer. An active strength test of the primary innervated muscle was performed for 3 s using a standardized procedure adapted from Mentiplay et al. The patient was instructed to press against the examiner's hand-and thus the hand-held dynamometer-as hard and as long as possible. The dynamometer recorded the strength and duration of the isometric contraction both graphically and numerically.
  The tested muscles included:
  L3: M. quadriceps femoris; L4: M. quadriceps femoris; M. tibialis anterior (TA); L5: M. TA; M. extensor hallucis longus (EHL); S1: M. gastrocnemius; M. triceps surae. Due to the small subgroups, the maximal isometric strengths of the quadriceps femoris muscle and triceps surae muscle were excluded from the analysis.The mean of the two closest of three values (N) was used for further analysis.
Time Frame: Baseline, 6 weeks, 6 months
Population: Maximal isometric strength was tested from the primary innervated muscle [L3: M. quadriceps femoris; L4: M. quadriceps femoris; M. tibialis anterior (TA); L5: M. TA; M. extensor hallucis longus (EHL); S1: M. gastrocnemius; M. triceps surae. Four patients missed the 6-month follow-up.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Newton
  M. tibialis anterior: Baseline: number analyzed (Participants) | 10
  M. tibialis anterior: Baseline | 91.5 (47.6)
  M. tibialis anterior: 6 weeks follow-up: number analyzed (Participants) | 10
  M. tibialis anterior: 6 weeks follow-up | 114.7 (71.8)
  M. tibialis anterior: 6 months follow-up: number analyzed (Participants) | 9
  M. tibialis anterior: 6 months follow-up | 142.0 (65.9)
  M. extensor hallucis longus: Baseline: number analyzed (Participants) | 9
  M. extensor hallucis longus: Baseline | 22.8 (9.0)
  M. extensor hallucis longus: 6 weeks follow-up: number analyzed (Participants) | 9
  M. extensor hallucis longus: 6 weeks follow-up | 34.3 (19.3)
  M. extensor hallucis longus: 6 months follow-up: number analyzed (Participants) | 7
  M. extensor hallucis longus: 6 months follow-up | 39.5 (12.6)

8. Primary Outcome: Changes in Nerve Tension Assessed by the Straight Leg Raising Test, Measured in Degrees
Description: Nerve tension of the affected spinal nerve root was assessed using the straight leg raise pain provocation test. A baseline bubble inclinometer was placed directly above the patella to measure the angle in degrees between the examination table and the elevated limb.
Time Frame: Baseline, 6 weeks, 6 months
Population: Four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Degree
  Baseline | 46.3 (23.4)
  6 weeks follow-up | 56.8 (17.0)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 66.3 (9.0)

9. Primary Outcome: Changes in Quality of Life Assessed by the Physical Component Summary of the 36-Item Short Form Health Survey
Description: General health was evaluated using the German version 2.0 of the 36-item Short Form Health Survey (SF-36). The PCS score aggregates four subscales-Physical Functioning, Role Physical, Bodily Pain, and General Health-into a standardized score ranging from 0 to 100, with higher scores reflecting better physical health.
Time Frame: Baseline, 6 weeks, 6 months
Population: Four patients missed the six-month follow-up. One participant failed to answer questions 4b-d of the SF-36 questionnaire at the six-week follow-up and questions 5b-c at both follow-ups, leading to missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
score on a scale
  Baseline | 35.2 (6.6)
  6 weeks follow-up: number analyzed (Participants) | 18
  6 weeks follow-up | 44.0 (8.2)
  6 months follow-up: number analyzed (Participants) | 14
  6 months follow-up | 51.7 (7.5)

10. Primary Outcome: Changes in Quality of Life Assessed by the Mental Component Summary of the 36-Item Short Form Health Survey
Description: General health was evaluated using the German version 2.0 of the 36-item Short Form Health Survey (SF-36). The MCS score aggregates four subscales-Vitality, Social Functioning, Role Emotional, and Mental Health-into a standardized score ranging from 0 to 100, with higher scores reflecting better mental health.
Time Frame: Baseline, 6 weeks, 6 months
Population: as for outcome 9
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
score on a scale
  Baseline | 44.2 (15.6)
  6 weeks follow-up | 53.8 (7.5)
  6 month follow-up: number analyzed (Participants) | 14
  6 month follow-up | 55.6 (4.3)

11. Primary Outcome: Changes in Physical Activity Assessed Using the International Physical Activity Questionnairee
Description: Physical activity was assessed using the self-administered short German version of the International Physical Activity Questionnaire (IPAQ) with a "last 7 days recall". Data were processed and analyzed according to the official IPAQ scoring protocol and reported in metabolic equivalents of task minutes per week
Time Frame: Baseline, 6 weeks, 6 months
Population: Four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: Metabolic equivalents of task-min./ week
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
Metabolic equivalents of task-min./ week
  Baseline | 2140.9 (2067.6)
  6 weeks follow-up | 2961.2 (2460.1)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 3718.0 (2846.5)

12. Primary Outcome: Changes in Disability According to the Oswestry Disability Index
Description: Disability was assessed using the German version of the Oswestry Disability Index. The ODI consists of 10 sections, each scored from 0 to 5. Scores are summed and expressed as a percentage ranging from 0 to 100, with higher scores indicating greater disability.
Time Frame: Baseline, 6 weeks, 6 months
Population: Four patients missed the six-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
Number analyzed (Participants) | 19
score on a scale
  Baseline | 37.2 (20.1)
  6 weeks follow-up | 16.7 (11.9)
  6 months follow-up: number analyzed (Participants) | 15
  6 months follow-up | 8.5 (12.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Lumbar Disc Herniation Associated With Radiculopathy
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03689400/Prot_SAP_000.pdf